CLINICAL TRIAL: NCT03062579
Title: Single-center, Open Label Trial of ACTEMRA® (Tocilizumab) as Monotherapy in Highly Active Neuromyelitis Optica Spectrum Disorders (NMOSD)
Brief Title: A Longitudinal Study of ACTEMRA® (Tocilizumab) as Monotherapy in Highly Active NMOSD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fu-Dong Shi (Other)
Responsible Party: Sponsor-Investigator, Fu-Dong Shi, Adjunct Professor of Neurology Department, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2017-YX-006
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Neuromyelitis Optica Spectrum Disorders; Neuromyelitis Optica; Devic's Disease
MeSH Terms: conditions — Neuromyelitis Optica | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ACTEMRA® (Tocilizumab) (Experimental): Tocilizumab will be intravenously administered as the dosage of 8 mg/kg every 4 weeks, 6 weeks if possible.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be intravenously administered as the dosage of 8 mg/kg every 4 weeks, 6 weeks if possible, without concurrent other immunosuppressive treatments.
  Other Names: ACTEMRA®

SUMMARY:
Neuromyelitis Optica Spectrum Disorder (NMOSD) is a severe inflammatory disease of the central nervous system characterized by relapsing optic neuritis and longitudinal extensive transverse myelitis. The specific autoantibody against aquaporin 4 (AQP4-ab) has been suggested to contribute to the pathogenesis of the disease. Peripheral blood plasma cells are a major source of AQP4-ab. Previous studies have observed increased IL-6 levels in serum and cerebrospinal fluid of patients with NMOSD, particularly during relapses. Exogenous interleukin (IL)-6 promotes the survival of plasma cells and their production of AQP4-ab in vitro. And blockade of IL-6 receptor signaling by an anti-IL-6 receptor antibody reduces the survival of plasma cells in vitro. Tocilizumab (ACTEMRA®), a humanized monoclonal antibody against the IL-6 receptor, has shown beneficial clinical effects in some patients with NMOSD when concomitant immunosuppressive medications were administered. However, the long-lasting biological effects of preceding immunotherapies such as rituximab might overlap with the subsequent tocilizumab therapy. To reduce the side effects of concomitant treatments to large extent and verify the beneficial effects of tocilizumab, we evaluate the safety and efficacy of tocilizumab as monotherapy in patients with NMOSD.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the drug tocilizumab as monotherapy contributes to reduce the average relapsing rate (ARR) and improve neurological disability in NMOSD patients, who still have experienced relapses when common immunosuppressive medications including rituximab had been used.

The primary (most important) objectives of this study are to determine: Whether bortezomib reduces relapse frequency in patients with relapsing NMO. The number of attacks during the one year treatment period will be compared to the number of attacks that occurred prior to initiation of tocilizumab treatment.

The secondary objectives are to determine:

The safety profile of tocilizumab in patients with NMO and whether tocilizumab improves walking, visual function and quality of life as measured by a variety of established disability scales.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of NMOSD, as defined by 2015 criteria.
2. NMOSD patients with at least one attack requiring rescue therapy in the last year or two attacks requiring rescue therapy in the last 2 years.
3. Provision of written informed consent to participate in the study.
4. Peripheral blood B cell count must be normal (5-20% of total lymphocytes) in subjects before administration of tocilizumab.
5. EDSS <= 7.5 (8 in special circumstances).

Exclusion Criteria:

1. Current evidence or known history of clinically significant infection (HSV, VZV, CMV, EBV, HIV, Hepatitis viruses, Syphilis, etc)
2. Pregnant, breastfeeding, or child-bearing potential during the course of the study
3. Patients will not participate in any other clinical therapeutic study or will not have participated in any other experimental treatment study within 30 days of screening
4. Participation in another interventional trial within the last 3 months
5. Heart or kidney insufficiency
6. Tumor disease currently or within last 5 years
7. Clinically relevant liver, kidney or bone marrow function disorder
8. Receipt of rituximab or any experimental B-cell depleting agent within 6 months prior screening and B-cells below the lower limit of normal.
9. Receipt of IVIG within 1 month prior to randomization.
10. Receipt of any other concomitant immunosuppressive therapies including corticosteroids, azathioprine, mycophenolate mofetil.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Median Number of Neuromyelitis Optica Spectrum Disorder (NMOSD) Attacks Per Year | Baseline, 12 months
  Compare annual relapses rate before and one year after initial tocilizumab administration

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Baseline, 12 months
  All adverse events and side effects related to this drug will be recorded.
Neurological Disability - Expanded Disability Scale Score (EDSS) | Baseline, 12 months
  The EDSS provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death.
Timed 25-foot Walk | Baseline, 12 months
  The Timed 25-Foot Walk test is a quantitative measure of lower extremity function. If required, the subject may use an appropriate assistive device to walk as quickly as he/she can from one end to the other end of a clearly marked, unobstructed, 25-foot course.
Change in Visual Acuity in eyes involved in NMOSD | Baseline, 12 months
  100% visual acuity and 2.5% contrast visual acuity are examined with high-contrast Sloan letter charts, which are readily available and provide a practical, quantitative, and standardized assessment of visual function. Each chart consists of rows of black letters (decreasing in size from top to bottom) on a white background.
Retinal Nerve Fiber Layer (RNFL) Thickness Determination | Baseline, 12 months
  Compared RNFL by use of Optical Coherence Tomography (OCT) before and one year after initial tocilizumab administration
Ganglion Cell Complex (GCC) Thickness Determination | Baseline, 12 months
  Compared GCC by use of Optical Coherence Tomography (OCT) before and one year after initial tocilizumab administration
Full Field Visual Evoked Response (VEP) P100 waves | Baseline, 12 months
  To determine the latency and amplitude of full field visual evoked response.
Number of new lesions by T2 hyperintensity in the spinal cord and brain MRI | Baseline, 12 months
  MRIs will be performed for standard of care purposes and will be used to evaluate imaging relapses. For this trial, the MRIs will be analyzed for counting the number of new lesions by T2 hyperintensity in the spinal cord and brain.
Counts of peripheral blood plasma cells | Baseline, 12 months
  Compare peripheral blood plasma cells before and one year after initial tocilizumab administration
Determination of serum immunoglobulins | Baseline, 12 months
  Compare immunoglobulins before and one year after initial tocilizumab administration

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Dong Shi, MD,PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No